CLINICAL TRIAL: NCT06133959
Title: Healthy ME: Advancing Health Equity in Lymphatic Pain and Lymphedema in Black and Hispanic Women With Breast Cancer
Acronym: HealthyME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2098673; RE33 (Other Grant/Funding Number: Oncology Nursing Foundation)
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: pain; lymphedema; breast cancer; behavior; intervention
MeSH Terms: conditions — Breast Neoplasms; Pain; Lymphedema; Behavior

STUDY DESIGN:
Intervention Model Description: Intervention and control arms
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will only know that they will be assigned to one of the two comparable behavioral and educational programs and they will not know which program is the intervention. Outcome assessors will not know the participants' assigned program throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-Lymph Control (Active Comparator): e-Lymph (Control). e-Lymph includes training sessions on the lymphatic system, lymphedema, lymphedema diagnosis and measurement, risk of lymphedema.
  Interventions: Behavioral: The-Optimal-Lymph-Flow (TOLF) Program
- The-Optimal-Lymph Flow (TOLF) Program (Experimental): TOLF includes training sessions on the lymphatic system, lymphedema, lymphedema diagnosis and measurement, risk of lymphedema, healthy diet, sleep hygiene, and daily lymphatic exercises. It has 8 avatar videos with step-by-step instructions for TOLF lymphatic exercises to promote lymph flow.
  Interventions: Behavioral: The-Optimal-Lymph-Flow (TOLF) Program

INTERVENTIONS:
Behavioral: The-Optimal-Lymph-Flow (TOLF) Program — TOLF includes training sessions on the lymphatic system, lymphedema, lymphedema diagnosis and measurement, risk of lymphedema, healthy diet, sleep hygiene, and daily lymphatic exercises. It has 8 avatar videos with step-by-step instructions for TOLF lymphatic exercises to promote lymph flow. It is expected that participants will complete initial in-person or telehealth virtual 40-minute session, and 3 virtual telehealth sessions with each session for 20-minute over the course of 8 weeks.

SUMMARY:
The goal of this two-phase project is to adapt The-Optimal-Lymph-Flow (TOLF) behavioral intervention to be culturally appropriate, and subsequently test the intervention in Black and Hispanic patients. The investigators have developed and tested behavioral intervention program TOLF that builds patients' self-management skills to promote lymph flow and results in complete pain reduction, reduced lymph fluid level, reversed mild lymphedema, and improved quality of life (QOL). Of concern, this promising intervention has not been adapted to reduce patient barriers (e.g., relevance, cost, time, travel, competing demands) and system barriers (e.g., intervention availability, staffing, therapist) to timely interventions faced by Black and Hispanic women. Specific aims are to:

Aim 1: Engage Black and Hispanic women (N=24) in adapting TOLF to be highly culturally appropriate. The investigators will conduct focus groups to refine TOLF focusing on barriers faced by and preferences of Black and Hispanic women.

Aim 2: Conduct a pilot randomized controlled trial (RCT) (N=60) equally allocating women to either 1) TOLF or 2) lymphedema education (e-Lymph) to examine feasibility, acceptability, and examine primary outcomes (lymphatic pain, pain severity and interference, and lymph fluid level) and secondary outcomes (daily living function, psychological distress, QOL, self-efficacy for pain management) of the culturally appropriate behavioral interventions.

DETAILED DESCRIPTION:
PURPOSE/SPECIFIC AIMS The purpose of this project is to adapt The-Optimal-Lymph-Flow (TOLF) behavioral intervention to be culturally appropriate, and subsequently test the intervention in Black and Hispanic patients. The investigators have developed and tested behavioral intervention program TOLF that builds patients' self-management skills to promote lymph flow and results in complete pain reduction, reduced lymph fluid level, reversed mild lymphedema, and improved quality of life (QOL). Of concern, this promising intervention has not been adapted to reduce patient barriers (e.g., relevance, cost, time, travel, competing demands) and system barriers (e.g., intervention availability, staffing, therapist) to timely interventions faced by Black and Hispanic women. Specific aims are to:

Aim 1: Engage Black and Hispanic women (N=24) in adapting TOLF to be highly culturally appropriate. The investigators will conduct focus groups to refine TOLF focusing on barriers faced by and preferences of Black and Hispanic women.

Aim 2: Conduct a pilot randomized controlled trial (RCT) (N=60) equally allocating women to either 1) TOLF or 2) lymphedema education (e-Lymph) to examine feasibility, acceptability, and examine primary outcomes (lymphatic pain, pain severity and interference, and lymph fluid level) and secondary outcomes (daily living function, psychological distress, QOL, self-efficacy for pain management) of the culturally appropriate behavioral interventions.

RATIONALE/SIGNIFICANCE OF THE STUDY. Lymphatic pain refers to pain, aching or soreness in the ipsilateral body or upper limb following breast cancer treatment. More than half of the 3.8 million women with breast cancer suffer lymphatic pain which leads to impaired daily living function, psychological distress, and compromised QOL. Most importantly, lymphatic pain is significantly associated with lymphedema, a chronic and incurable condition caused by an abnormal accumulation of lymph fluid. Black and Hispanic women are three times as likely to suffer from lymphedema compared to White women. Timely intervention for lymphatic pain can decrease the risk and severity of lymphedema. However, there are persistent barriers to timely interventions faced by Black and Hispanic women with breast cancer - a group at high risk for developing lymphedema, pain, and other negative breast cancer related outcomes.

THEORETICAL FRAMEWORK. Self-efficacy theory guides the project. Behavioral pain interventions focus on training patients on self-management skills to be implemented in their daily lives.

MAIN RESEARCH VARIABLES. Behavioral pain intervention (IV), Outcomes (DVs): lymphatic pain, pain severity and interference, lymph fluid level, daily living function, psychological distress, QOL, self-efficacy for pain management.

DESIGN. Qualitative and randomized clinical trial (RCT)

SETTING. All participants will be recruited from UMKC University Health and surrounding communities.

SAMPLES. Black and Hispanic women with lymphatic pain

METHODS. Focus groups will be conducted with Black and Hispanic women to gather data that will lead to culturally appropriate adaptation of TOLF. Then, a pilot RCT will be used to examine feasibility, acceptability, and evidence of future efficacy of this culturally adapted intervention.

IMPLICATIONS FOR PRACTICE. The successful completion of the project will advance health equity in pain and lymphedema by making this culturally appropriate, highly accessible, and effective behavioral intervention available to Black and Hispanic women.

ELIGIBILITY:
Inclusion Criteria:

* The participants are Black and Hispanic women (over age 18) with lymphatic pain following breast cancer treatment. These women will be recruited for the Phase I focus groups (N=24), and the Phase II RCT (N=60). Participants will include women who 1) have received surgical treatment for breast cancer at least 3 months prior to the study enrollment, 2) report persistent or intermittent pain/aching/soreness in the ipsilateral body or upper limb; 3) self-identify as either Black or Hispanic; and 4) are able to understand the study protocols presented in English.

Exclusion Criteria:

* Exclusion criteria include: 1) presence of a serious psychiatric condition (e.g., schizophrenia, suicidal intent) indicated by medical chart, treating oncologist or other staff, or study staff interactions that would contraindicate safe study participation; 2) known metastatic disease (Stage IV), recurrence of cancer, or lymphedema due to cancer recurrence, or other bulk disease in the thoracic or cervical regions; 3) were diagnosed or treated for lymphedema.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Lymphatic Pain | Pre-intervention (0 week) and Post-intervention (13 week)
  The Breast Cancer and Lymphedema Symptom Experience Index (BCLE-SEI) Part I, a reliable and valid self-report instrument, is used to assess self-reported lymphatic pain, i.e., aching or soreness or tenderness.
Pain Severity and Interference | Pre-intervention (0 week) and Post-intervention (13 week)
  Brief Pain Inventory-Short Form (BPI-SF) will be used to measure pain severity and interference. The measure demonstrated reliability and validity.65 The BPI-SF consists of four items assessing pain severity (worst, least, average, and current pain) and seven items assessing pain interference in the past week.

SECONDARY OUTCOMES:
Lymph Fluid Level | Pre-intervention (0 week) and Post-intervention (13 week)
  A bioelectrical impedance analysis (BIA) device is used to assess lymph fluid level. The device measures the resistance of the extracellular fluid (i.e. the impedance) in terms of the fluid ratio, taking into consideration the ratio between the dominant and non-dominant arms.
Daily Living Function: | Pre-intervention (0 week) and Post-intervention (13 week)
  The Breast Cancer and Lymphedema Symptom Experience Index (BCLE-SEI) Part II is used to measure activity of daily living (ADLs). The 13-item subscale of ADLs in BCLE-SEI Part II is used to assess self-reported difficulty in performing thirteen ADLs.
Psychological Distress | Pre-intervention (0 week) and Post-intervention (13 week)
  The 12-item subscale of psychological/emotional distress subscale from the BCLE-SEI Part II is used to assess the distress of being frustrated, sad, guilt/self-blame, worried, irritable, fearful, angry, lonely, helpless, hopeless, anxious, and depressed. Cronbach's alpha for the psychological/emotional distress subscale was 0.91.
Patients' Quality of life | Pre-intervention (0 week) and Post-intervention (13 week)
  Global Health Scale (PROMIS GHS) is used to measure quality of life (QOL) captures self-perception of QOL on a scale from 1 (poor), 2 (fair), 3 (good), 4 (very good) to 5 (excellent). This tool has good reliability (a= 0.80-0.86).
Self-efficacy for Pain Management | Pre-intervention (0 week) and Post-intervention (13 week)
  The 5-item Chronic Pain Self-Efficacy Scale81 with good reliability69-70 is used to assess patients' certainty about their degree of pain control, pain during daily activities, controlling pain during sleep, and making pain reductions without extra medication.

CONTACTS AND LOCATIONS:
Overall Officials: Mei R Fu, Principal Investigator — University of Missouri, Kansas City
Locations (1):
- University of Missouri-Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
We will not share any individual participant data during and after study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT06133959/Prot_SAP_000.pdf